CLINICAL TRIAL: NCT02784405
Title: Safety and Effectiveness of the Self-aPposing, bAlloon-delivered, dRug-eluting Stent for the Treatment of the Coronary Artery Disease: A multiCenter Registry
Brief Title: Self-apposing Stentys Stents Registry
Acronym: SPARTA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Claudio Moretti, MD, A.O.U. Città della Salute e della Scienza
Other Study IDs: sparta2016
Record Dates: First submitted 2016-04-22; First posted 2016-05-27 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Coronary Artery Disease
Keywords: percutaneous coronary intervention; stent implantation
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
Self-apposing, drug-eluting Stentys coronary stents represent a valuable tool for the treatment of coronary artery stenosis. Their ability to adapt to widely varying vessel calibers and to auto-expand after their release to self-appose to vessel walls is particularly useful in the presence of ectasic coronary arteries or significant vessel tapering. The investigators planned this study to assess the feasibility, the effectiveness and the safety of the implantation of self-apposing, drug-eluting Stentys stents for percutaneous coronary intervention.

Consecutive patients undergoing percutaneous coronary intervention with implantation of a self-apposing Stentys stent were enrolled in this multi center registry. Inclusion criteria were age ≥ 18 years and ability to provide informed consent. No exclusion criteria were defined.

Primary end-point of the study is the occurrence of MACE (death, myocardial infarction, stent thrombosis, unplanned hospitalization for unstable angina, target lesion revascularization). Secondary end-points include individual components of MACE, procedural complications (periprocedural MI, bleedings, access site complication, failure to cross stent struts with guidewire in the treatment of bifurcation, failure to delivery the stent, contrast-induced nephropathy), bleedings at follow up.

DETAILED DESCRIPTION:
Rationale: Choice of the appropriate size of stents in the treatment of coronary artery stenosis can often be challenging. Marked tapering of vessels' diameter in their proximal-distal development may lead to sub-optimal results. Distal under-expansion of the drug-eluting stent (DES) or vessel perforation may occur if a larger DES, best suited for the proximal diameter, is chosen. Proximal DES under-sizing with struts malapposition may happen if a smaller DES, fitting the distal diameter, is implanted. Moreover, ectasic vessels present irregular and varying diameter, which may lead as well to segmental malapposition or under-expansion of DES. Self-apposing stents can overcome these limitations thanks to their ability to self-expand also after their release in the vessel and to adapt to a wide range of vessel diameters. Multiple generation of self-apposing, drug-eluting stents have been developed, with progressive amendments pertaining the stent-deployment technique (from deployment by covering-sheath retraction to balloon-delivery) and the drug released (from paclitaxel to sirolimus). The last generation of the self-apposing stents is represented by the sirolimus-eluting, balloon-delivered Xposition S stents. Studies assessing performance of this stent are however limited in sample size and length of follow up, and are mainly controlled trials. Few data are available regarding the clinical outcomes of the self-apposing Stentys stents in a "real-life" setting.

Aim of this study is to assess the feasibility, the effectiveness and the safety of the implantation of self-apposing, drug-eluting Stentys stents for percutaneous coronary intervention.

Study population: Patients undergoing percutaneous coronary intervention with implantation of a self-apposing Stentys stent.

Primary analysis: Longitudinal cohort follow up

Study end-points:

Primary efficacy end-point:

* Major adverse cardiovascular events (MACE) (a composite end point including death, myocardial infarction (MI, excluding periprocedural MI), stent thrombosis, unplanned hospitalization for unstable angina, target lesion revascularization (TLR))

Secondary efficacy end-points:

* Individual components of MACE (death, MI, stent thrombosis, unplanned hospitalization, TLR)

Secondary safety end-points:

* Procedural complications:

  * Periprocedural MI
  * Bleedings
  * Access site complication
  * Failure to cross stent struts with guidewire in the treatment of bifurcation
  * Failure to delivery the stent
  * Contrast-induced nephropathy
* Bleedings at follow up

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* ability to provide informed consent

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients undergoing percutaneous treatment of coronary artery disease with implantation of a self-apposing, drug-eluting, Stentys stent
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events (MACE) | 12 months
  A composite end-point of death, myocardial infarction, stent thrombosis, unplanned hospitalization for unstable angina, target lesion revascularization

SECONDARY OUTCOMES:
Death | 12 months
Myocardial Infarction | 12 months
  Incident rate of myocardial infarction
Stent thrombosis | 12 months
  Incident rate of stent thrombosis
Target lesion revascularization | 12 months
  Incident rate of target lesion revascularization
Unplanned hospitalization for unstable angina | 12 months
  Incident rate of unplanned hospitalization for unstable angina
Procedural and in-hospital complications | 30 days
  Incident rate of periprocedural myocardial infarction, bleedings and access site complication, failure to cross stent struts with guidewire in the treatment of bifurcation, failure to delivery the stent, contrast-induced nephropathy
Bleeding events | 12 months
  Incident rate of bleedings classified according to the BARC criteria

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Moretti, MD, Principal Investigator — Division of Cardiology, Department of Medical Sciences, AO Città della Salute e della Scienza, University of Turin, Turin, Italy; Antonio Montefusco, MD, Principal Investigator — Division of Cardiology, Department of Medical Sciences, AO Città della Salute e della Scienza, University of Turin, Turin, Italy; Bernardo Cortese, MD, Principal Investigator — Interventional Cardiology, A.O. Fatebenefratelli Milano, Italy
Locations (14):
- Italy (12):
  - Division of Cardiology, Mazzoni Hospital, Ascoli Piceno
  - Ferrarotto Hospital, University of Catania, Catania
  - Division of Cardiology, ASL TO4, Cirié
  - Division of Cardiology, Santa Maria dei Battuti Hospital, Conegliano
  - Division of Cardiology, Ospedale Civile di Legnano - ASST Ovest Mi, Legnano
  - Interventional Cardiology, Azienda Ospedaliera Fatebenefratelli, Milan
  - Division of Cardiology, Federico II University, Napoli
  - Division of Cardiology, Santa Corona Hospital, Pietra Ligure
  - Division of Cardiology, Fondazione Toscana G Monasterio, Pisa
  - Division of Cardiology, Policlinico Umberto I, La Sapienza University, Roma
  - Division of Cardiology, ASST Bergamo Ovest, Treviglio
  - AO Città della Salute e della Scienza, Turin
- Cardiology Department, Manipal Klang Hospital, Kuala Selangor, Malaysia
- Division of Cardiology, Medical University of Silesia, Katowice, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lu H, IJsselmuiden AJ, Grundeken MJ, Nassif M, de Vries AG, Weevers A, Scholte M, Spaargaren R, Wykrzykowska JJ, Tijssen JG, de Winter RJ, Koch KT. First-in-man evaluation of the novel balloon delivery system STENTYS Xposition S for the self-apposing coronary artery stent: impact on longitudinal geographic miss during stenting. EuroIntervention. 2016 Mar;11(12):1341-5. doi: 10.4244/EIJY15M05_07. PMID 25983027
- [Background] Pyxaras SA, Schmitz T, Naber CK. The STENTYS Self-Apposing(R) stent. EuroIntervention. 2015;11 Suppl V:V147-8. doi: 10.4244/EIJV11SVA34. No abstract available. PMID 25983152
- [Background] Farooq V, Gomez-Lara J, Brugaletta S, Gogas BD, Garcia-Garcia HM, Onuma Y, van Geuns RJ, Bartorelli A, Whitbourn R, Abizaid A, Serruys PW. Proximal and distal maximal luminal diameters as a guide to appropriate deployment of the ABSORB everolimus-eluting bioresorbable vascular scaffold: a sub-study of the ABSORB Cohort B and the on-going ABSORB EXTEND Single Arm Study. Catheter Cardiovasc Interv. 2012 May 1;79(6):880-8. doi: 10.1002/ccd.23177. Epub 2011 Oct 5. PMID 22514149
- [Background] Uren NG, Schwarzacher SP, Metz JA, Lee DP, Honda Y, Yeung AC, Fitzgerald PJ, Yock PG; POST Registry Investigators. Predictors and outcomes of stent thrombosis: an intravascular ultrasound registry. Eur Heart J. 2002 Jan;23(2):124-32. doi: 10.1053/euhj.2001.2707. PMID 11785994
- [Background] Yew KL, Kang Z. First-in-man unprotected left main stenting with Stentys Xposition S self-apposing sirolimus eluting stent and optical coherence tomography guidance: The emerging panacea for left main intervention. Int J Cardiol. 2015 Dec 15;201:628-30. doi: 10.1016/j.ijcard.2015.08.035. Epub 2015 Aug 4. No abstract available. PMID 26340130
- [Background] Buccheri D, Orrego PS, Cortese B. Drug-eluting stent treatment of left main coronary artery disease: the case for a sirolimus-eluting, autoexpandable alternative. An optical coherence tomography analysis. Int J Cardiol. 2015 Nov 15;199:119-20. doi: 10.1016/j.ijcard.2015.07.006. Epub 2015 Jul 11. No abstract available. PMID 26188831
- [Background] van Geuns RJ, Yetgin T, La Manna A, Tamburino C, Souteyrand G, Motreff P, Koch KT, Vrolix M, IJsselmuiden A, Amoroso G, Berland J, Montalescot G, Teiger E, Christiansen EH, Spaargaren R, Wijns W. STENTYS Self-Apposing sirolimus-eluting stent in ST-segment elevation myocardial infarction: results from the randomised APPOSITION IV trial. EuroIntervention. 2016 Feb;11(11):e1267-74. doi: 10.4244/EIJV11I11A248. PMID 26865444
- [Background] Yew KL. Longitudinal stent foreshortening of Stentys Xposition S self-apposing stents and its impact on overlapping stenting strategy. Int J Cardiol. 2016 Feb 1;204:187-8. doi: 10.1016/j.ijcard.2015.11.176. Epub 2015 Nov 25. No abstract available. PMID 26666346
- [Derived] Montefusco A, D'Ascenzo F, Gili S, Smolka G, Chieffo A, Baumbach A, Escaned J, Sganzerla P, Tomassini F, Secco GG, Ugo F, Tamburino C, Nicolino A, Mancone M, Poli A, Yew KL, Cirillo P, Wanha W, Pastormerlo LE, di Summa R, Sardella G, Colombo A, Gaita F, Cortese B. Self-expandable sirolimus-eluting stents compared to second-generation drug-eluting stents for the treatment of the left main: A propensity score analysis from the SPARTA and the FAILS-2 registries. Catheter Cardiovasc Interv. 2019 Feb 1;93(2):208-215. doi: 10.1002/ccd.27809. Epub 2018 Oct 8. PMID 30298593